CLINICAL TRIAL: NCT07219602
Title: A Placebo-Controlled, Double-Blind, Randomized, Phase 3 Study to Evaluate the Effect of Obicetrapib 10 mg and Ezetimibe 10 mg Fixed-Dose Combination or Obicetrapib 10 mg Daily on Top of Guideline-Recommended Lipid-Lowering Therapy in Participants With Type 2 Diabetes and/or Metabolic Syndrome (RUBENS Trial)
Brief Title: A Study to Evaluate the Effect of Obicetrapib/Ezetimibe 10 mg Fixed-Dose Combination or Obicetrapib 10 mg Daily on Top of Guideline-Recommended Lipid-Lowering Therapy in Participants With Type 2 Diabetes and/or Metabolic Syndrome
Acronym: RUBENS
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: NewAmsterdam Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: OBEZ-303
Record Dates: First submitted 2025-10-20; First posted 2025-10-22 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Lipidemia; Type 2 Diabetes (T2DM); Metabolic Syndrome (MetS)
MeSH Terms: conditions — Hyperlipidemias; Diabetes Mellitus, Type 2; Metabolic Syndrome | interventions — Ezetimibe

STUDY DESIGN:
Intervention Model Description: This protocol includes a 12-week, 3-arm, placebo-controlled, double-blind treatment section, followed by a 40-week open-label extension period. All patients receive the FDC of obicetrapib 10mg and ezetimibe 10 mg, regardless of the intervention received in the double-blind treatment section of this trial.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Obicetrapib/Ezetimibe (Experimental): obicetrapib 10 mg + ezetimibe 10 mg FDC daily
  Interventions: Drug: obicetrapib 10 mg + ezetimibe 10 mg FDC daily
- Obicetrapib (Experimental): obicetrapib 10 mg daily
  Interventions: Drug: Obicetrapib 10 mg
- Placebo (Placebo Comparator): Placebo on top of guideline-recommended lipid-lowering therapy
  Interventions: Other: Placebo
- Open-Label Extension (Experimental): Open-Label Extension (OLE) with the FDC of Obicetrapib 10 mg and Ezetimibe 10 mg
  Interventions: Drug: obicetrapib 10 mg + ezetimibe 10 mg FDC daily

INTERVENTIONS:
Drug: obicetrapib 10 mg + ezetimibe 10 mg FDC daily — FDC
  Arms: Obicetrapib/Ezetimibe; Open-Label Extension
Drug: Obicetrapib 10 mg — monotherapy
  Arms: Obicetrapib
Other: Placebo — placebo on top of guideline-recommended lipid modifying therapy
  Arms: Placebo

SUMMARY:
This study will be a placebo-controlled, double-blind, randomized, Phase 3 study to evaluate the efficacy, safety, and tolerability of obicetrapib 10 mg, both as a fixed-dose combination (FDC) with ezetimibe 10 mg and as monotherapy, on top of guideline-recommended lipid-lowering therapy in patients with metabolic syndrome and/or Type 2 Diabetes Mellitus.

ELIGIBILITY:
Inclusion Criteria:

* fasting serum LDL-C ≥ 70 mg/dL (≥1.81 mmol/L)
* Have fasting TG ≥150 mg/dL (≥1.7 mmol/L) and <400 mg/dL (<4.5 mmol/L)
* Know diagnosis of T2DM OR have metabolic syndrome defined as fasting TG ≥150 mg/dL (≥1.7mmol/L) and <400 mg/dL (<4.5 mmol/L) and at least 2 risk factors
* Are on stable guideline-recommended lipid-lowering therapy
* Estimated glomerular filtration rate ≥15 mL/min/1.73 m2

Exclusion Criteria:

* Have current or any previous history of New York Heart Association class III or IV heart failure or left ventricular ejection fraction <30%
* Have been hospitalized for heart failure within 5 years prior to Screening
* Have uncontrolled severe hypertension
* Have a formal diagnosis of homozygous familial hypercholesterolemia
* HbA1c ≥10.0% (≥0.100 hemoglobin fraction) or a fasting glucose ≥270 mg/dL (≥15.0 mmol/L) at Screening
* active liver disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2028-03 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
The percent change from Baseline to Day 84 in LDL-C compared with placebo for the following treatment groups: - obicetrapib 10 mg + ezetimibe 10 mg FDC treatment group; and - obicetrapib 10 mg monotherapy treatment group | 84 days

SECONDARY OUTCOMES:
Percent change from Baseline to Day 84 in non-HDL-C for the obicetrapib 10 mg + ezetimibe 10 mg FDC treatment group compared with the placebo group | Day 84
Percent change from Baseline to Day 84 in HDL-C for the obicetrapib 10 mg + ezetimibe 10 mg FDC treatment group compared with the placebo group | 84 days
Percent change from Baseline to Day 84 in ApoB for the obicetrapib 10 mg + ezetimibe 10 mg FDC treatment group compared with the placebo group | 84 days
Percent change from Baseline to Day 84 in ApoA1 for the obicetrapib 10 mg + ezetimibe 10 mg FDC treatment group compared with the placebo group | 84 days
Percent change from Baseline to Day 84 in non-HDL-C for the obicetrapib 10 mg monotherapy treatment group compared with the placebo group; | 84 days
Percent change from Baseline to Day 84 in HDL-C for the obicetrapib 10 mg monotherapy treatment group compared with the placebo group | Day 84
Percent change from Baseline to Day 84 in ApoB for the obicetrapib 10 mg monotherapy treatment group compared with the placebo group | Day 84
Percent change from Baseline to Day 84 in ApoA1 for the obicetrapib 10 mg monotherapy treatment group compared with the placebo group | Day 84
Percent change from Baseline to Day 84 in lipoprotein (a) (Lp[a]) for the obicetrapib 10 mg + ezetimibe 10 mg FDC treatment group compared with the placebo group | Day 84
Percent change from Baseline to Day 84 in Lp(a) for the obicetrapib 10 mg monotherapy treatment group compared with the placebo group | Day 84

OTHER OUTCOMES:
Percent change from Baseline over time in LDL-C | 40 weeks
  The percent change from Baseline at every visit for LDL-C
Proportion of participants that achieve LDL-C <100 mg/dL (<2.6 mmol/L), LDL-C <70 mg/dL (<1.8 mmol/L), and LDL-C <55 mg/dL (<1.4 mmol/L) | 40 weeks
  The percent change from Baseline at every visit in the proportion of participants that achieve LDL-C <100 mg/dL (<2.6 mmol/L), LDL-C <70 mg/dL (<1.8 mmol/L), and LDL-C <55 mg/dL (<1.4 mmol/L)
Percent change from Baseline over time in non-HDL-C | 40 weeks
  The percent change from Baseline at every visit for non-HDL-C
Percent change from Baseline over time in ApoB | 40 weeks
  The percent change from Baseline at every visit in ApoB
Percent change from Baseline over time in total cholesterol | 40 weeks
  The percent change from Baseline at every visit for total cholesterol
Percent change from Baseline over time in triglycerides | 40 weeks
  The percent change from baseline at every visit for triglycerides
Percent change from Baseline over time in HDL-C | 40 weeks
  the percent change from Baseline at every visit for HDL-C
Percent change from Baseline over time in Lp(a) | 40 weeks
  the percent change from Baseline at every visit for Lp(a)

IPD SHARING:
Plan to Share IPD: Yes